CLINICAL TRIAL: NCT06702085
Title: Effects of Lifestyle Changes on Tinnitus in Older Adults With Metabolic Syndrome
Brief Title: Lifestyle Changes in Older Adults With Metabolic Syndrome and Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer, Department of Physical Therapy for Cardiovascular/Respiratory Disorders and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004623
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Tinnitus; Metabolic Syndrome X; Obesity; Elderly; Weight Loss
MeSH Terms: conditions — Tinnitus; Metabolic Syndrome; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (Experimental): thirty older adults (with obesity, metabolic syndrome, and chronic subjective tinnitus) administered supervised changes in their lifestyle (walking exercise for 40 minutes applied on treadmill for three time per week and low caloric diet) for twelve weeks
  Interventions: Behavioral: Lifestyle Management
- second group (No Intervention): thirty older adults (with obesity, metabolic syndrome, and chronic subjective tinnitus) served as control patients who did not receive any changes in their lifestyle

INTERVENTIONS:
Behavioral: Lifestyle Management — patients administered supervised changes in their lifestyle (walking exercise for 40 minutes applied on treadmill for three time per week and low caloric diet) for twelve weeks
  Arms: first group

SUMMARY:
The problem of tinnitus (subjective type) is prevalent in obese older adults with different diseases such as metabolic syndrome. The changes of lifestyle are very important to lose weight, improve tinnitus and metabolic syndrome

DETAILED DESCRIPTION:
Sixty older adults (with metabolic syndrome with chronic subjective tinnitus) with obesity were selected in a equal random manner to be classified into the first group that administered changes in their lifestyle (exercise applied on treadmill and low caloric diet) for twelve successive weeks and second group that was not administered lifestyle changes

ELIGIBILITY:
Inclusion Criteria:

* obese person (class one obesity)
* patients with metabolic syndrome
* patients with chronic subjective tinnitus (bilateral complaint from more than six months).
* older adults aging 65 years and more
* both sexes will be included

Exclusion Criteria:

* respiratory insult
* cardiac insult
* liver insult
* kidney insult
* lower limb insult
* neurological insult

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-identified gender identity
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale of tinnitus severity | twelve weeks
  it is scale (10 cm) that will assess severity of tinnitus

SECONDARY OUTCOMES:
visual analogue scale of tinnitus related discomfort | twelve weeks
  it is a scale (10 cm) that will assess tinnitus related discomfort
tinnitus handicap inventory | twelve weeks
  it is a questionnaire that will assess quality of life in tinnitus population
body mass index | twelve weeks
  it will be assessed at morning after evacuation of bowel and bladder
waist circumference | twelve weeks
  it will be measured at the level of umbilicus
triglycerides | twelve weeks
  it will be measured in the serum
high density lipoprotein | twelve weeks
  it will be assessed in the serum
systolic blood pressure | twelve weeks
  it will be assessed by mercury sphygmomnameter
diastolic blood pressure | twelve weeks
  it will be assessed by mercury sphygmomnameter
fasting blood glucose | twelve weeks
  it will be measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, Lecturer, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University, Dokki, Giza Governorate
  - faculty of physical therapy Cairo university, Dokki, Giza Governorate

REFERENCES:
- [Derived] Ismail AMA, Tolba AMN. Effectiveness of lifestyle-modification approach (a randomized-controlled program of diet restriction and treadmill walking exercise) on elderly's metabolic syndrome-associated subjective tinnitus. Eur Arch Otorhinolaryngol. 2025 Aug;282(8):4307-4315. doi: 10.1007/s00405-025-09494-7. Epub 2025 Jun 11. PMID 40500514